CLINICAL TRIAL: NCT07202767
Title: Intraocular Lens Calculation Using Artificial Intelligence
Status: Not yet recruiting | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-015
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Cataract
Keywords: cataract; lens diameter; artificial intelligence
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Cohort with MRI: Patients who are included in this study who additionally receive a cerebral MRI
  Interventions: Device: Swept-Source Anterior Segment OCT
- Study cohort without MRI: Study cohort who doesn't receive an MRI
  Interventions: Device: Swept-Source Anterior Segment OCT

INTERVENTIONS:
Device: Swept-Source Anterior Segment OCT — Device: Swept-Source Anterior Segment OCT The CASIA-2 (Tomey, Japan) is a high-resolution swept-source anterior segment OCT with CE certification. The device allows for incomplete visualization of the lens, including the anterior and posterior lens curvature.
  Device: AS-OCT + Placido disc corneal topography The MS-39 (CSO, Italy) is a non-invasive device that combines Placido topography with OCT-based anterior segment tomography.
  Device: Wave-front abberomtery The OSIRIS aberrometer is a standard tool for examining corneal aberration and measuring the ocular wavefront.
  Device: Swept-Source OCT The IOLMaster 700 (Carl Zeiss Meditec, Germany) is a standard swept-source OCT used for eye examinations.
  Device: AS-OCT The ANTERION (Heidelberg Engineering, Germany) is an anterior segment swept-source OCT.
  Diagnostic Test: Refraction Subjective Refraction evaluation using the cross-cylinder method

SUMMARY:
The aim of this study is to investigate the lens diameter (LD) as a useful parameter in intraocular lens (IOL) power calculation by using several different non-invasive imaging techniques. The aim is to establish an accurate model for lens diameter estimation and subsequently evaluate the influence of the LD on the effective postoperative lens position. The comparability of the different devices in terms of variability between the biometric measurements will also be assessed.

By then combining these two approaches with artificial intelligence, the aim is to develop a new approach to effectively incorporate the LD in IOL power calculation and improve patient's outcome in the long run.

DETAILED DESCRIPTION:
During uncomplicated cataract operation, the clouded natural lens is being removed and replaced with an artificial intraocular lens (IOL). To achieve optimal postoperative outcomes for patients, the power of the implanted artificial lens is calculated prior to surgery.

Significant progress has been made in calculation concepts over the past 20 years, including the introduction of regression, vergence and ray tracing. More recently, approaches incorporating artificial intelligence have emerged.

All these formulae are based on the biometric data of the eye. This includes parameters such as axial eye length, corneal curvature, central corneal thickness, anterior chamber depth and the refractive indices of the eye's optical segments. By including all these variables, modern formulas aim to deliver the best possible postoperative outcomes.

One variable that has not been included in the calculation thus far is the diameter of the natural lens. Large parts of the lens are covered by the iris. Even with medically dilated pupils the peripheral parts cannot be visualized, and subsequently not adequately reproduced using established imaging methods. This has made implementation in IOL power calculation difficult.

In everyday clinical practice, however, anterior segment OCT imaging devices are equipped with features that allow for an estimation of lens diameter. This is achieved by extrapolating the anterior and posterior curvature of the natural lens, which unfortunately makes this approach prone to error. Other imaging techniques, such as magnetic resonance imaging, are impractical in routine clinical practice due to time and cost considerations. However, they could be highly beneficial for future predictive approaches of the lens diameter The aim of this study is to develop a model for incorporating the lens diameter into IOL calculation. This will be achieved by using different imaging technologies to determine the actual lens diameter. The diameter will then be predicted using available biometric variables.

ELIGIBILITY:
Inclusion criteria

* age 21 years and older
* planned uncomplicated bilateral cataract surgery
* availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits
* ability to consent to the participation in the study
* signed informed consent

Exclusion criteria

* multifocal IOL
* combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* PEX, previous ocular surgery, severe trauma or any pathology that could lead to an unstable capsular bag
* glaucoma or any other retinal disease that may affect visual acuity significantly
* pregnancy
* pre-operative visual acuity below 0.1 Snellen decimal (1.0 Log MAR)
* pupil diameter <4mm

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected at Kepler University Clinic Linz at the Departement of Ophthalmology and Optometry.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Prediction model to estimate lens diameter with different measurement tools (swept-AS segment OCT; anterior segment-OCT and Placido topography with OCT-based anterior segment tomography; wave-front abberometry; swept-source OCT and optical biometer) | preoperatively, 4 and 12 weeks post cataract surgery
  Developing a prediction model to accurately estimate the lens diameter using biometric parameters (swept-source anterior segment Optical Coherence Topography (Casia-2), Placido topography combined with Optical Coherenece Topography-based anterior segment tomography (MS-39), wave-front abberometry (OSIRIS), Swept-Source Optical Coherence Tomography (IOLMaster 700) and anterior segment swept-source OCT (Anterion).
Prediction model to estimate lens diameter with cerebral Magnetic Resonance Imaging | 12 weeks post cataract surgery
  Developing a prediction model to accurately estimate the lens diameter using cerebral Magnetic Resonance Imaging to examine ocular configuration

SECONDARY OUTCOMES:
IOL calculation concept an artificial intelligence approach | preoperatively, 4 and 12 weeks post cataract surgery
  Development of a new IOL calculation concept which includes the lens diameter using an artificial intelligence approach
Different measurement modalities for the biometry of the eye | 4 and 12 weeks post cataract surgery
  Comparison of different measurement modalities (swept-source anterior segment Optical Coherence Topography; anterior segment-Optical Coherence Tomography and Placido topography with Optical Coherenece Topography-based anterior segment tomography; wave-front abberometry; swept-source Optical Coherence Tomography and optical biometer) for the biometry of the eye

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD PhD, Principal Investigator — JKU Linz
Locations (1):
- Kepler University Clinic, Linz, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided